CLINICAL TRIAL: NCT05104034
Title: Comprehensive Risk Assessment and Prevention Plan of Osteoporosis and Sarcopenia for the Elderly Participating in Community-based Long-term Care Services
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 202106076RIND
Record Dates: First submitted 2021-10-11; First posted 2021-11-02 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2023-09

CONDITIONS: Osteoporosis; Sarcopenia; Frailty
Keywords: Osteoporosis; Sarcopenia; Quality of life; Intrinsic capacity; Frailty
MeSH Terms: conditions — Osteoporosis; Sarcopenia; Frailty | interventions — Therapeutics; Health Services Needs and Demand; Exercise; Nutritional Status; Pharmaceutical Services

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Screening group (Experimental): Inform the elderly about the results of the screening and recommend those with moderate to high risk of fracture to receive active examination and treatment.
  Interventions: Behavioral: Osteoporosis screening and treatment as needed
- Multi-component integrated intervention (Experimental): Introduce integrated services of health education, nutrition, rehabilitation, pharmaceutical care, and other multi-specialties to assist study participants with health promotion
  Interventions: Behavioral: Osteoporosis screening and treatment as needed; Behavioral: Sarcopenia; Behavioral: Exercise; Dietary Supplement: Nutrition; Behavioral: Pharmaceutical care
- Delayed intervention (Placebo Comparator): receive general care after collecting basic information, and provide health education related information such as osteoporosis sarcopenia. After two year's follow-up, multi-disciplinary team intervention service will be implemented.
  Interventions: Behavioral: Osteoporosis screening and treatment as needed

INTERVENTIONS:
Behavioral: Osteoporosis screening and treatment as needed — All residents underwent screening using the Fracture Risk Assessment Tool (FRAX) and Mobile dual-energy X-ray absorptiometry (DXA) (Horizon Wi, Hologic Inc., Bedford, MA). Our study nurses actively assisted osteoporosis treatment if indicated.
Behavioral: Sarcopenia — Sarcopenia assessment adhered to the 2019 Consensus Update on Sarcopenia Diagnosis and Treatment by the Asian Working Group for Sarcopenia guideline. Following screening, individuals identified with sarcopenia underwent tailored interventions involving exercise and nutrition as deemed necessary.
  Arms: Multi-component integrated intervention
Behavioral: Exercise — TheraBand (resistance band) was utilized as the exercise tool within the community. T
  Arms: Multi-component integrated intervention
Dietary Supplement: Nutrition — Nutrition Nutritional education programs aim to increase protein food serving and the choice of those with insufficient dietary intake. Protein supplement was added if indicated.
  Arms: Multi-component integrated intervention
Behavioral: Pharmaceutical care — We collected drug information of the elderly. Detailed and real-time prescription drug information was retrieved from the National Health Insurance PharmaCloud System. A pharmaceutical care team performed patient-centered drug review and discussion every three to six months.
  Arms: Multi-component integrated intervention

SUMMARY:
The purpose of this project is:

1. Provide the epidemiological data of the prevalence, incidence, and risk factors of osteoporosis and sarcopenia among the elderly in rural areas.
2. Screen osteoporosis and sarcopenia among the elderly and provide with assistance for following care in order to improve the diagnosis and treatment rates of osteoporosis and sarcopenia
3. Construct a pragmatic and integrated care service model for osteoporosis and sarcopenia in the elderly people from rural areas

DETAILED DESCRIPTION:
Detailed Description:

Investigators plan to use a stepped-wedge cluster randomized trial that allocates participants into the following three groups:

1. Screening group: Inform the elderly about the results of the screening and recommend those with moderate to high risk of fracture to receive active examination and treatment.
2. Multi-disciplinary team intervention group: Introduce integrated services of health education, nutrition, rehabilitation, medication evaluation and other multi-specialties to assist study participants with health promotion.
3. Control group (Delayed intervention): receive general care after collecting basic information, and provide health education related information such as osteoporosis sarcopenia. After two year's follow-up, multi-disciplinary team intervention service will be implemented.

ELIGIBILITY:
Inclusion Criteria:

* Age≥ 50 old and lived in the community

Exclusion Criteria:

* Life expectancy less than two years

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-09-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The changes of Quality of life and quality adjusted life year | one year, two year, 3 year, four year
  Using EQ5D / WHOQOL Brief questionnaires to measure quality of life and evaluate the changes after intervention. In addition, to calculate quality adjusted life year by using utility index derived from qualify of life measurement.
Intrinsic capacity | one year, two year, 3 year, four year
  To define if the Intrinsic capacity would be changed after intervention
Institutionalilzation rate | one year, two year, 3 year, four year
  To define if the Institutionalilzation rate would be changed after intervention

SECONDARY OUTCOMES:
Incidence of fall | one year, two year, 3 year, four year
  To define if the fall frequency would be changed after intervention
Incidence of fracture | one year, two year, 3 year, four year
  To define if the incidence of fracture would be changed after intervention
Incidence of unexpected hospitalization | one year, two year, 3 year, four year
  To define if the unexpected hospitalization would be changed after intervention

OTHER OUTCOMES:
Incidence of mortality | one year, two year, 3 year, four year
  To define if the Incidence of mortality would be changed after intervention
Changes of drug related problems | one year, two year, 3 year, four year
  Under the assumption of the intervention of pharmaceutical care in the multi-component group can improve the DRPs of the elderly, we also measured the changes of drug number, anticholinergic burden and adherence (using the Adherence to Refills and Medications Scale).
Phyiscal performance | one year, two years
  Changes of muscle strength, body composition, physical performance, activites of daily living
Sarcopenia related outcomes | one year, two years
  We follow sarcopenia diagnosis rate, treatment rate, changes of muscle mass, fat, and muscle-fat index
Osteoporosis related outcomes | one year, two years
  We follow osteoporosis diagnosis rate, treatment rate, adherence to osteoporosis treatment, and changes of bone mineral density
Mental health | one year, two years
  We use Geriatric Depression Scale and Chinese Happiness Inventory to measure depression and happiness
Nutrition related outcomes | one year, two years
  Changes in protein intake, dietary/caloric intake, nutritional status
Cognition | one year, two years
  Changes in MMSE

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Yunlin branch, Douliu, Yunlin County, Taiwan

REFERENCES:
- [Derived] Fu SH, Lai WJ, Yen HK, Kukreti S, Li CY, Hung CC, Wang CY. Addressing healthcare disparities and improving osteoporosis management in rural communities: a cluster randomized control trial. Arch Osteoporos. 2025 Jan 28;20(1):15. doi: 10.1007/s11657-025-01498-4. PMID 39875677